CLINICAL TRIAL: NCT02851264
Title: Diagnostic Value of Virtual Chromoendoscopy With Optical Enhancement Technology in Early Esophageal Squamous Neoplasia: A Prospective Comparative Study
Brief Title: Diagnostic Value of Optical Enhancement Technology in Early Esophageal Squamous Neoplasia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2016SDU-QILU-10
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Early Esophageal Squamous Neoplasia
Keywords: Early Esophageal Squamous Neoplasia; optical enhancement technology; virtual chromoendoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — According to virtual chromoendoscopy with optical enhancement technology and Lugol iodine chromoendoscopy ,endoscopic biopsies will be taken at suspicious lesions respectively .
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Optical enhancement technology examination: After routine examination by white-light endoscopy,the imaging mode will be switched to optical enhancement.Suspicious area will be recorded in detail. Then all enrolled patients will have their esophagus sprayed with iodine solution. Suspicious area will be also recorded in detail.After that biopsy specimens will be obtained respectively by forceps from each suspicious lesion recorded for histologic diagnosis.

SUMMARY:
The aims of the present study：

1. To investigate the diagnosing value of optical enhancement technology for early esophageal squamous neoplasia.
2. To assess the detection rate of early esophageal squamous neoplasia by virtual chromoendoscopy with optical enhancement technology .

DETAILED DESCRIPTION:
Detection and differentiation of esophageal squamous neoplasia (ESN) are of value in improving patient outcomes.Optical enhancement technology can serves in the diagnosis of GI neoplasia. However, its performance in ESN has not yet been reported.The aims of the present study is:

1. To investigate the diagnosing value of optical enhancement technology for early esophageal squamous neoplasia.
2. To assess the detection rate of early esophageal squamous neoplasia by virtual chromoendoscopy with optical enhancement technology .

ELIGIBILITY:
Inclusion Criteria:

1. Patients with high-risk factors for esophageal squamous cell carcinoma who meet any of follows：

   * Long term living in the high incidence area of esophageal squamous cell carcinoma ；
   * First degree relatives have a history of esophageal squamous cell carcinoma ；
   * Previous history of esophageal lesions （ esophageal squamous neoplasia ）；
   * The patients having a history of cancer；
   * A long history of smoking ；
   * A long history of drinking ；
   * Having bad eating habits such as eating fast, hot diet, high salt diet, eating pickles.
2. Patients aged between 40 to 74 years old.

Exclusion Criteria:

1. Having advanced esophageal carcinoma;
2. After esophageal surgery or endoscopic treatment ;
3. Known esophageal radiotherapy or chemotherapy ;
4. Esophageal stenosis;
5. Acute bleeding;
6. A known allergy to iodine;
7. Coagulopathy (prothrombin time <50% of control, partial thromboplastin time >50 seconds);
8. Having food retention;
9. Severe hepatic ,renal, cardiovascular or metabolic dysfunction ;
10. Being pregnant or lactating;

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients screened that fulfill the eligibility criteria at Qilu Hospital, Shandong University will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The detection rate of early esophageal squamous neoplasia by optical enhancement technology. | 12 months
  The detection rate of early esophageal squamous neoplasia by using optical enhancement and Lugol chromoendoscopy.

SECONDARY OUTCOMES:
The diagnostic accuracy of optical enhancement technology on early esophageal squamous neoplasia. | 12 months
  Patients will be prospectively recruited to evaluate the diagnostic sensitivity, specificity and accuracy of early esophageal squamous neoplasia by using optical enhancement and Lugol chromoendoscopy.
The different rate of adverse events between optical enhancement and Lugol chromoendoscopy. | 12 months
The observation time of optical enhancement and Lugol chromoendoscopy. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China